CLINICAL TRIAL: NCT01319890
Title: The 'SILVERMAN1' Trial Single Incision Laparoscopic Versus Existing Resection (Minimal Access) for Neoplasia
Acronym: SILVERMAN 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Irish Clinical Outcomes in Research and Education (Network)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: Silverman1
Record Dates: First submitted 2011-03-02; First posted 2011-03-22 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Right Colon Tumors
Keywords: all histologic subtypes; benign; malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Right Colectomy for colonic tumors: The group of patients enrolled will be patients with biopsy proven right colon tumors, both benign and malignant. These patients will then be subdivided into those having conventional laparoscopic right colectomy and SILS right colectomy
  Interventions: Procedure: Patients will be divided in two groups- those having right colectomy by standard laparoscopy and those having Single Incision Laparoscopic Surgery (SILS)

INTERVENTIONS:
Procedure: Patients will be divided in two groups- those having right colectomy by standard laparoscopy and those having Single Incision Laparoscopic Surgery (SILS) — Patients will be divided into 2 arms- those with right colon tumors treated by conventional laparoscopic right colectomy and those having a Single Incision Laparoscopic Surgery (SILS)

SUMMARY:
Current evidence regarding the optimal surgical approach to potentially curable right colonic cancer is based on numerous, well designed randomised controlled clinical trials. Currently, eminence based opinion suggests that an alternative surgical technique, single incision laparoscopic surgery (SILS), may improve short and long term outcomes after minimally invasive right colonic resection. A true, prospective analysis comparing standard of care (laparoscopic right hemicolectomy) and this "new" therapy(SILS) has yet to be published. Having established the optimum treatment modality the minimally invasive approach to right colonic tumors the results will be communicated at national and international meetings.

DETAILED DESCRIPTION:
The 'SILVERMAN' 1 Trial Single Incision Laparoscopic Versus Existing Resection (Minimal Access) for Neoplasia- A Multi-institutional Randomised Controlled Trial

Applicant:

Professor Desmond C Winter, Institute for Clinical Outcomes Research and Education (iCORE), St. Vincent's University Hospital, Elm Park, Dublin 4, Ireland.

winterd@indigo.ie

Background Colonic cancer is the third commonest cause of cancer mortality in women and men in the developed world[1]. Old age, adenomatous colorectal polyps, inflammatory bowel disease, low intake of dietary fibre and family history of colorectal cancer all predispose to the development of colonic cancer[2-4]. Certain genetic syndromes such as Hereditary Non-Polyposis Colon Cancer (HNPCC), Familial Adenomatous Polyposis (FAP), Peutz-Jeghers Syndrome (PJS) and Juvenile Polyposis have a significant lifetime risk of developing colonic cancer[5-8]. Historically, open surgery has been the mainstay of treatment for localised, potentially curable colonic cancer. Laterally, minimally invasive or laparoscopic surgery has largely supplanted open surgery in the management of colonic cancer[9,10,11]. Published data have shown that laparoscopic assisted resection has equivalent oncological outcomes in terms of long term survival when compared to conventional open surgery. Similarly, Level 1 evidence from the major randomised controlled trials in this field suggests that laparoscopic colonic resection confers advantages over the open approach during the perioperative period in terms of reduced requirement for parenteral narcotics and oral analgesics, earlier restoration of intestinal function, earlier ambulation, and shorter hospital stay. To date there remains no consensus or accepted guidelines on the surgical management of potentially curable right colonic cancer. The NHS published guidelines on management of colorectal cancer simply state that surgeons offering their patients potentially curative laparoscopic resections should be appropriately trained in such specialist techniques12. Currently, surgeons competent in minimal access surgery favour laparoscopic right hemicolectomy as the technique of choice for right colonic resection. Intestinal continuity can be restored intracorporeally, or extracorporeally by exteriorising the mobilised segment of ileum/right and transverse colon.

The advent of "single incision laparoscopic surgery" (SILS) has further advanced the minimally invasive approach to the management of complex surgical diseases. SILS, currently in the embryonic stages of development, utilises a single incision to insert a single access device into the abdominal cavity under direct vision. Typically, the device is inserted in the midline and utilises a 2-3cm incision around the umbilicus, itself an embryonic natural orifice.

The optical and operating trocars are inserted through the access device and the procedure is carried out as a conventional laparoscopic procedure. Many short case series and reports have been published describing the feasibility of SILS in performing complex surgical procedures for both benign and malignant disease[13,14,15]. Specialised, complex colorectal procedures such as proctocolectomy with ileal pouch-anal anastomosis (IPAA), ileocolic resection for terminal ileal Crohn's mass and colonic resection for cancer have been successfully performed using single incision laparoscopic surgery[16,17,18,19]. To date, several short series of SILS right hemicolectomy have been published in the literature[20,21].Thus, rather than a new or novel technique, SILS is a derivation of laparoscopic surgery, performed through a single incision. There is no evidence in the literature that SILS colectomy confers any disadvantages over conventional laparoscopic surgery and to dtae, there are no reports of SILS putting patients at increased risk of complication. Postulated benefits of SILS colectomy over conventional laparoscopic colectomy include reduced number of incisions, improved cosmesis, less pain, faster return to normal activities/work and shorter hospital stay. Heretofore, there has been no randomised controlled clinical trial comparing SILS and standard laparoscopic right hemicolectomy for cancer. Having previously demonstrated the benefits of laparoscopic resection over open resection in the treatment of colon cancer we feel the time is ripe to further extrapolate these data by comparing laparoscopic right hemicolectomy with a proposed new treatment modality, single incision laparoscopic right hemicolectomy, in the format of a multicentre, international randomised controlled clinical trial.

Knowledge transfer/implementation Current evidence regarding the optimal surgical approach to potentially curable right colonic cancer is based on numerous, well designed randomised controlled clinical trials. Currently, eminence based opinion suggests that an alternative surgical technique, SILS, may improve short and long term outcomes after minimally invasive right colonic resection. A true, prospective analysis comparing standard of care (laparoscopic right hemicolectomy) and this "new" therapy(SILS) has yet to be published. Having established the optimum treatment modality the minimally invasive approach to right colonic tumors the results will be communicated at national and international meetings. Findings will be submitted to an international surgical journal to ensure maximal communication of results and will be made available to national and international academic societies to enable the establishment of guidelines of best practice for surgical management of right colonic cancer.

Objective

To compare patient outcome following standard of care (laparoscopic right hemicolectomy) and an alternative, established, recognized therapy (SILS right hemicolectomy) for the treatment of right colonic tumors. Specific research questions include:

1. Which treatment modality confers least perioperative morbidity and mortality in the surgical management of right colonic tumors?
2. Does treatment influence length of time to discharge home and return to activities of daily living?
3. Are treatment modalities equivalent in terms of extent of resection (lymph node yield, resection margins etc)?

Strategy An Irish based, multi-centre, international trial will be performed with the aim of comparing two treatment modalities for patients presenting with right colonic cancer. Pre-operative details, intraoperative findings and post-operative course will be prospectively accrued by the operating surgeon. Each surgeon has previous experience in performing this procedure and currently offer SILS colectomy to their patients outside of a clinical trial setting. All patients will be followed up and primary and secondary end-points will be recorded.

Primary End-points

1. Qualitative - Lymph node yield

   * Histopathological grade of specimen
   * Conversion rate
   * 30 day mortality
   * Cancer free survival

   Secondary Endpoints
2. Quantitative- operative time

   * pain scores (visual analog scale)
   * cosmesis satisfaction
   * earlymorbiditywound/respiratory /urosepsis, thromboembolic,cardiorespiratory, anastomotic leak, intra- abdominal abscess and reoperation
   * Intravenous narcotic/ oral analgesic requirements
   * Resumption of intestinal function/ diet
   * Duration to discharge home
   * Return to normal activity

Study Design The study will be an international multi-centred ,randomized controlled trial. Ethical approval will be sought prior to study implementation.

Inclusion criteria

1. Age 18-85 years
2. Histologic confirmation of right colonic cancer
3. Informed consent

Exclusion criteria

1. Inability to give informed consent (e.g. dementia)
2. Previous midline laparotomy incision
3. T4 tumour diagnosed on pre-operative imaging or intra-operatively
4. Previous pelvic irradiation
5. FAP/ HNPCC
6. Colonic carcinoma against a background of ulcerative colitis.
7. Emergent surgery for perforated/obstructing right colonic cancer

Study outline All patients with histologically confirmed right colonic tumours will be eligible for the study. Individual patient consent will be sought. Each patient will be randomized at the pre-operative visit the day prior to surgery; thus, each patient will know, in advance, which procedure they are undergoing.

Patients should be staged pre-operatively with Computed Tomography of abdomen and pelvis to facilitate therapeutic and operative strategy. All patients will be given prophylaxis against deep vein thrombosis (sequential intermittent pneumatic compression devices/compression stockings and low molecular weight heparin).

A single, prophylactic dose of antibiotics will be given perioperatively; the choice of antibiotic will be determined according to institutional guidelines. Operative procedure will be according to standard practice.

At laparoscopic right hemicolectomy, pneumoperitoneum will be established following insertion of a 12mm umbilical port. Two or 3 further operating trocars (5mm) will be inserted; the number and position will be at the operating surgeons discretion. When it is necessary to use more than two 5mm trocars to complete the procedure this will be recorded. Ligation of the vascular pedicle must be performed intracorporeally using an endovascular stapling device, endoclips or an electrothermal coagulation device. If the major vessels are ligated extracorporeally when the mobilised colon has been exteriorised for resection the procedure will be classified as "laparoscopic assisted"- i.e. converted to an open procedure- for the purposes of this trial. Intestinal continuity will be restored extracorporeally using end to end, end-to side or side-to side anastomosis. The type of anastomosis will be at the surgeons' discretion (stapled vs. handsewn) and will be recorded.

Patients having SILS right hemicolectomy will receive the same perioperative care as those undergoing conventional laparoscopic resection. The SILS access device is inserted through a 4-5cm incision (max 6cm incision), 2cm above and 1 cm below the umbilicus. The access device utilises three 5mm trocars facilitating entry to the peritoneal cavity. The choice of access device will be at individual surgeons' discretion. In the event of additional ports being required to complete a SILS minimally invasive procedure the number of additional trocars used will be recorded. Oral fluids will be commenced on the evening of surgery and diet will be introduced the following morning, depending on clinical status. Urinary catheters will be removed on post-operative day 1 and ambulation encouraged.

Data Collection Data collection will be performed by the operating surgeon, a designated member of the surgical team (present at time of operation) or Dr. Martin, Co-PI on the study, and recorded on an electronic pro-forma and submitted to an on-line database (the iCore website- Institute for Clinical Outcomes in Research and Education). Each patient enrolled in the study will be given a study number and all data will be registered under this number. Patients will thus be deidentified. Any data that could potentially identify patients such as D.O.B/ date of surgery, date of discharge will be excluded . It will include patient demographics (age, sex), American Society of Anaesthesiologists (ASA) grade and specific co-morbidities, intervention performed, operation performed, number of ports used, technique for ligation of vascular pedicle, type of anastomosis, re-intervention during index admission (radiological or operative) in-hospital morbidity (myocardial infarction, deep vein thrombosis, pulmonary embolism, wound infection, abscess requiring drainage, urosepsis, renal failure or respiratory insufficiency), mortality, analgesic requirements, time to return to diet, time to discharge to home. Further details will be recorded at post-operative visits including the number of days alive following discharge, reinterventions within 12 months and patient satisfaction. Each patient will be seen at 3 and 12 months post-operatively. For those patients from out of state who prefer to be followed up locally we will perform a telephone interview at the timelines outlined. Patient satisfaction will be determined using the Short Form (SF-36) questionnaire at 3 and 12 months.

Sample Size The main short-term endpoints of the study are both qualitative (lymph node yield, grade of specimen) and quantitative (operative time, cosmesis satisfaction, resumption of normal diet/intestinal function, length of hospital stay). Cancer-related survival is the main long-term primary end-point. The working hypothesis is that there will be no significant differences in this variable between SILS and conventional laparoscopic right hemicolectomy, but that differences in variables related to the short-term outcome (i.e. morbidity and duration of hospital stay) would favour SILS. We assume that a difference in cancer-related survival of less than 15% between treatments indicates an equivalent efficacy. Assuming a 70% 5-year cancer-related survival in the laparoscopic colectomy group, a minimum of 100 patients per group is required to show that both surgical techniques are equivalent with an α level of 0•20 and a β error of 0•05. Recruitment of patients is not expected to be difficult because evidence to date is convincing of at least equivalent outcome and we believe that most patients would hope to be assigned to the SILS group, with potentially shorter hospital stay, less pain and improved cosmesis. From a surgeon's perspective, SILS is technically feasible and represents only a slight modification of the conventional laparoscopic procedure.

Hospital Inclusion and Patient Accrual All eligible patients (see exclusion criteria) presenting to participating hospitals with right colonic tumors will be recruited for the trial. . Each patient will be randomized at the pre-operative visit the day prior to surgery; thus, each patient will know, in advance, which procedure they are undergoing.

Patients will be furnished with a patient information leaflet and will have the implications of inclusion in the trial explained to them by the operating surgeon. It will be explained that non-willingness to participate in the trial will not have any negative impact on their treatment. If the patient is willing to participate in the trial, verbal and written consent will be obtained prior to transfer to the operating theatre.

Randomisation schedules will be in blocks, with the proposed treatment delivered in writing in sequentially numbered, opaque, sealed envelopes. If inferiority of efficacy is demonstrable on preliminary statistical analysis, the trial will be stopped prematurely to prevent harm to patients. We aim to perform a preliminary analysis of the pooled data at 6/12/18/24 months or when 100/150/200 patients have been entered into the trial; whichever comes first will prompt preliminary analysis. Each adverse event will be included in the electronic file of each patient in the study. The data will then be communicated with the PI at each site participating in the study. In the event of one technique being of greater risk to patients, the lead center in Dublin, Ireland will terminate the study prematurely. Similarly, in the event of a PI in the study being unhappy with the outcomes of the study, they are free to withdraw from the trial at any time. This withdrawal will be reported in publishing the data.

Statistical Analysis Data will be assessed according to the intention-to-treat principle. Because the scope of the study is non-metastatic colon cancer, patients in whom metastases are detected intra-operatively will not be included in the analyses of long-term outcome. Survival is calculated from surgical resection of primary tumour to the last visit or death. For cancer-related survival, patients who die from other causes will be censored from the study at time of death. Probability curves will be constructed with the Kaplan-Meier method and compared with the log-rank test.

We will use proportional-hazards modeling with forward selection to determine the influence of patients' baseline characteristics on cancer-related survival and other variables. The surgical procedure and any variable reaching a p value of less than 0•10 in the univariate analysis will then undergo multivariate analysis to identify independent predictors.

Categorical variables will be compared by χ2 test, with the Yates correction when necessary. Continuous variables will be compared by the Student's t test or the Mann-Whitney U test, depending on their distribution.

All p values will be two-sided with a p value of less than 0•05 indicating a significant difference. All calculations will be performed with SPSS (version 18.0 for Windows).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years
2. Histologic confirmation of right colonic cancer
3. Informed consent

Exclusion Criteria:

1. Inability to give informed consent (e.g. dementia)
2. Previous midline laparotomy incision
3. T4 tumour diagnosed on pre-operative imaging or intra-operatively
4. Previous pelvic irradiation
5. FAP/ HNPCC
6. Colonic carcinoma against a background of ulcerative colitis.
7. Emergent surgery for perforated/obstructing right colonic cancer
8. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven right colon tumors, benign and malignant, aged 18-85 years will be included.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
operative time | Within 3 months of surgery
  The length of time taken to complete each procedure will be recorded
pain scores (visual analog scale) | Within 90 days of surgery
  Pain scores will be calculated on day 1,2 and 3 post-operatively and on first clinic visit
cosmesis satisfaction | within 1 year of surgery
Peri-operative complications will be recorded within 3 months of the index operation | within 3 months of surgery
  early morbidity- wound/respiratory / urinary sepsis, thromboembolic, cardiorespiratory, anastomotic leak, intra-abdominal abscess, reoperation
Intravenous narcotic/ oral analgesic requirements | Within 3 months of surgery
  Patients analgesic requirements will be calculated both in-hospital and after discharge records will be detailed at clinic visit
Resumption of intestinal function/ diet - Duration to discharge home - Return to normal activity | within 3 months of surgery
  Time to passage of flatus, bowel motion and dietary intake will be recorded while the patient is in hospital
Duration to discharge home | within 3 months of date of surgery
  Time patient is in hospital will be recorded on discharge from the unit
Return to normal activity/work | within 6 months of surgery
  The timeframe from surgery to resumption of normal activities of daily living and return to work will be determined at patients second clinic visit

SECONDARY OUTCOMES:
Lymph node yield | within 3 months of surgery
  The pathology specimen detailing the lymph node count will be entered at first clinic visit post-operatively or within 3 months of surgery
Conversion rate | Within 3 months of surgery
  The conversion from a laparoscopic to an open procedure will be known at time of operation and will be recorded prior to patient discharge or at the first clinic visit
30 day mortality | within 3 months of surgery
  Mortality rates within 30 days will be recorded during the hospitl stay or within 3 months of surgery
Cancer free survival | 5 years following the date of surgery
  Cancer free survival will be determined at 5 years from the index surgery. Expected 5 years, disease free survival should be equivalent if the hypothesis is true.

CONTACTS AND LOCATIONS:
Overall Officials: Des Winter, MD FRCSI, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (1):
- St. Vincent's University Hospital, Dublin, Ireland

REFERENCES:
- [Background] MACDOUGALL IP. THE CANCER RISK IN ULCERATIVE COLITIS. Lancet. 1964 Sep 26;2(7361):655-8. doi: 10.1016/s0140-6736(64)92474-2. No abstract available. PMID 14188905
- [Background] SEER Cancer Statistics Review, 1975-2007, National Cancer Institute. Bethesda, MD, http://seer.cancer.gov/csr/1975_2007/
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Burkitt DP, Walker AR, Painter NS. Effect of dietary fibre on stools and the transit-times, and its role in the causation of disease. Lancet. 1972 Dec 30;2(7792):1408-12. doi: 10.1016/s0140-6736(72)92974-1. No abstract available. PMID 4118696
- [Background] Cannon-Albright LA, Skolnick MH, Bishop DT, Lee RG, Burt RW. Common inheritance of susceptibility to colonic adenomatous polyps and associated colorectal cancers. N Engl J Med. 1988 Sep 1;319(9):533-7. doi: 10.1056/NEJM198809013190902. PMID 2841598
- [Background] Vogelstein B, Fearon ER, Hamilton SR, Kern SE, Preisinger AC, Leppert M, Nakamura Y, White R, Smits AM, Bos JL. Genetic alterations during colorectal-tumor development. N Engl J Med. 1988 Sep 1;319(9):525-32. doi: 10.1056/NEJM198809013190901. PMID 2841597
- [Background] Kinzler KW, Nilbert MC, Su LK, Vogelstein B, Bryan TM, Levy DB, Smith KJ, Preisinger AC, Hedge P, McKechnie D, et al. Identification of FAP locus genes from chromosome 5q21. Science. 1991 Aug 9;253(5020):661-5. doi: 10.1126/science.1651562.
- [Background] Resta N, Simone C, Mareni C, Montera M, Gentile M, Susca F, Gristina R, Pozzi S, Bertario L, Bufo P, Carlomagno N, Ingrosso M, Rossini FP, Tenconi R, Guanti G. STK11 mutations in Peutz-Jeghers syndrome and sporadic colon cancer. Cancer Res. 1998 Nov 1;58(21):4799-801. PMID 9809980
- [Background] Lacy AM, Garcia-Valdecasas JC, Delgado S, Castells A, Taura P, Pique JM, Visa J. Laparoscopy-assisted colectomy versus open colectomy for treatment of non-metastatic colon cancer: a randomised trial. Lancet. 2002 Jun 29;359(9325):2224-9. doi: 10.1016/S0140-6736(02)09290-5. PMID 12103285
- [Background] Clinical Outcomes of Surgical Therapy Study Group; Nelson H, Sargent DJ, Wieand HS, Fleshman J, Anvari M, Stryker SJ, Beart RW Jr, Hellinger M, Flanagan R Jr, Peters W, Ota D. A comparison of laparoscopically assisted and open colectomy for colon cancer. N Engl J Med. 2004 May 13;350(20):2050-9. doi: 10.1056/NEJMoa032651. PMID 15141043
- [Background] Guillou PJ, Quirke P, Thorpe H, Walker J, Jayne DG, Smith AM, Heath RM, Brown JM; MRC CLASICC trial group. Short-term endpoints of conventional versus laparoscopic-assisted surgery in patients with colorectal cancer (MRC CLASICC trial): multicentre, randomised controlled trial. Lancet. 2005 May 14-20;365(9472):1718-26. doi: 10.1016/S0140-6736(05)66545-2. PMID 15894098
- [Background] http://www.acpgbi.org.uk/assets/documents/COLO_guides.pdf
- [Background] Kim HJ, Lee JI, Lee YS, Lee IK, Park JH, Lee SK, Kang WK, Cho HM, You YK, Oh ST. Single-port transumbilical laparoscopic appendectomy: 43 consecutive cases. Surg Endosc. 2010 Nov;24(11):2765-9. doi: 10.1007/s00464-010-1043-9. Epub 2010 Apr 16. PMID 20396909
- [Background] Podolsky ER, Curcillo PG 2nd. Single port access (SPA) surgery--a 24-month experience. J Gastrointest Surg. 2010 May;14(5):759-67. doi: 10.1007/s11605-009-1081-6. Epub 2010 Feb 13. PMID 20155330
- [Background] Elsey JK, Feliciano DV. Initial experience with single-incision laparoscopic cholecystectomy. J Am Coll Surg. 2010 May;210(5):620-4, 624-6. doi: 10.1016/j.jamcollsurg.2009.12.030. PMID 20421017
- [Background] Geisler DP, Condon ET, Remzi FH. Single incision laparoscopic total proctocolectomy with ileopouch anal anastomosis. Colorectal Dis. 2010 Sep;12(9):941-3. doi: 10.1111/j.1463-1318.2009.02115.x. Epub 2009 Nov 6. PMID 19895601
- [Background] Heeney A, O'Connor DB, Martin S, Winter DC. Single-port access laparoscopic surgery for complex Crohn's disease. Inflamm Bowel Dis. 2010 Aug;16(8):1273-4. doi: 10.1002/ibd.21163. No abstract available. PMID 19902539
- [Background] Remzi FH, Kirat HT, Geisler DP. Laparoscopic single-port colectomy for sigmoid cancer. Tech Coloproctol. 2010 Sep;14(3):253-5. doi: 10.1007/s10151-009-0545-8. Epub 2009 Dec 2. PMID 19953288
- [Background] Uematsu D, Akiyama G, Matsuura M, Hotta K. Single-access laparoscopic colectomy with a novel multiport device in sigmoid colectomy for colon cancer. Dis Colon Rectum. 2010 Apr;53(4):496-501. doi: 10.1007/DCR.0b013e3181ce677a. PMID 20305452
- [Background] Ramos-Valadez DI, Patel CB, Ragupathi M, Bartley Pickron T, Haas EM. Single-incision laparoscopic right hemicolectomy: safety and feasibility in a series of consecutive cases. Surg Endosc. 2010 Oct;24(10):2613-6. doi: 10.1007/s00464-010-1017-y. Epub 2010 Apr 3. PMID 20364353
- [Background] Boni L, Dionigi G, Cassinotti E, Di Giuseppe M, Diurni M, Rausei S, Cantore F, Dionigi R. Single incision laparoscopic right colectomy. Surg Endosc. 2010 Dec;24(12):3233-6. doi: 10.1007/s00464-010-1100-4. Epub 2010 May 13. PMID 20464415